CLINICAL TRIAL: NCT00498693
Title: Hypoxia Inducible factor1-Alpha Genetic Polymorphism of Obstructive Sleep Apnea
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Peilin Lee, National Taiwan University Hospital
Other Study IDs: 9561701013
Record Dates: First submitted 2007-07-08; First posted 2007-07-10 (Estimated); Last update posted 2009-01-14 (Estimated); Status verified 2009-01

CONDITIONS: Sleep Apnea, Obstructive
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Specific Aim

1. To identify specific SNPs of HIF-1 gene related to cardiovascular disease in OSA patients (CVD-OSA)
2. To assay the functional activity of high risk SNPs of HIF-1 on the transcription of VEGF gene
3. To confirm that the serum level of VEGF in CVD-OSA patients with high risk SNPs of HIF-1 are higher than CVD-OSA patients without

DETAILED DESCRIPTION:
Obstructive sleep apnea syndrome(OSAS) is characterized with recurrent collapse of upper airway during sleep and results in hypoxia and sleep fragmentation. The repeated episodes of hypoxia and sympathetic hyperactivity result in cardiovascular complications, including atherosclerosis, hypertension, coronary artery disease and heart failure. Our data showed among 309 consecutively-admitted OSA patients, 54% patients had cardiovascular diseases.

The hypoxia in OSA is characterized as chronic and intermittent, which leads to sophisticated adaptive mechanisms, like activations of transcriptional factors and critical signaling pathways. HIF-1 is a central component of transcriptional factors involved in hypoxia-induced transcription of specific genes. There are two subunits of HIF-1 transcription factor, which interact with the consensus hypoxia response element in the target genes. The HIF-1 alpha activity is regulated by proline hydroxylation modification and ubiquitination, which is oxygen-tension dependent. HIF-1 alpha target genes encode proteins that increase oxygen delivery, such as vascular endothelial growth factor(VEGF). Our oligo-microarray study showed both HIF and VEGF expression in OSA patients was 1.3 times of control group, which decreased to 46% and 57% respectively after one-month CPAP treatment.

HIF-1 alpha polymorphism could result in increased HIF-1 alpha activity and microvessel density. In clinical observation, HIF-1 polymorphism has been reported to be associated with high altitude adaptation, formation of coronary collaterals in CAD and phenotype of cancer. These findings were possibly explained with effect of HIF on modulation of VEGF.

Several genetic polymorphisms were reported to be associated with OSA, which included TNF alpha, angiotensin converting enzyme and haptoglobin. Only hepatoglobin phenotype is proved to be a risk factor for cardiovascular disease in OSA. In most studies, the patient number is less than suggested.

Therefore, in this study, we hypothesized that HIF-1 gene polymorphism was associated with cardiovascular disease in OSA. And by using large-scale of study population(1000 OSA patients), we examined all regions of the HIF-1 alpha to detect single-nucleotide polymorphisms(SNPs), evaluated the pattern of linkage disequilibrium to compose haplotypes in the gene, and performed association studies in OSA patients with and without cardiovascular disease to achieve the following 3 objectives:(1)To identify specific SNPs of HIF-1 alpha gene related to cardiovascular disease in OSA patients (CVD-OSA).(2)To assay the functional activity of high risk SNPs of HIF-1 alpha on the transcription of VEGF gene.(3)To confirm that the serum level of VEGF in CVD-OSA patients with high risk SNPs of HIF-1 are higher than CVD-OSA patients without. The findings are expected to stratify the risk of OSA patients to specific outcome, or response to specific therapy.

ELIGIBILITY:
Inclusion Criteria:

* Severe obstructive sleep apnea (AHI>=30/hr) age, sex, BMI match control subject

Exclusion Criteria:

* Patients were excluded when: (1) refused to participate in this study, (2) had severe obstructive pulmonary disease or active neurological events, (3) enrolled in other studies at the same time

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients referred sleep center to rule out obstructive sleep apnea
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2006-03

CONTACTS AND LOCATIONS:
Overall Officials: Hey-Dong Wu, M.D., Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan Univeristy Hospital, Taipei, Taiwan

REFERENCES:
- [Derived] Pandit JJ. Structure-function relationships: a breath of fresh air--or just more hot air--in sleep apnoea research? Respiration. 2008;76(1):16-8. doi: 10.1159/000127578. Epub 2008 May 8. No abstract available. PMID 18583924